CLINICAL TRIAL: NCT04350723
Title: Awake Prone Position in Hypoxemic Patients With Coronavirus Disease 19 (COVI-PRONE): A Randomized Clinical Trial
Brief Title: Awake Prone Position in Hypoxemic Patients With Coronavirus Disease 19 COVID-19 (COVI-PRONE)
Acronym: COVI-PRONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: King Abdullah International Medical Research Center (Other); McMaster University (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Waleed Al-Hazzani, Principal Investigator, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2154
Record Dates: First submitted 2020-04-14; First posted 2020-04-17 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Corona Virus Infection; Covid19; COVID-19
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Intervention Model Description: A multicenter, parallel-group randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Awake Proning (Experimental): The oxygen mask or NIPPV or HFNC will be initiated at the treating team's discretion. The patient will be observed for 15 minutes to ensure that: SPO2 > 90% and the patient is tolerating oxygen mask or NIPPV or HFNC treatment.
  Once the patient achieves the above parameters within 15 minutes of initiating oxygen therapy through any modality, the healthcare team will start awake proning.
  Interventions: Procedure: Awake Proning
- Control - Standard of Care (No Intervention): The patient will receive usual care without proning at the discretion of the treating team.
  The oxygen mask or NIPPV or HFNC will be initiated, the choice of starting oxygen mask versus NIPPV versus HFNC will be up to the treating team, the patient will be observed for 15 minutes to ensure that: SPO2 > 90% and the patient is tolerating NIPPV or HFNC treatment.

INTERVENTIONS:
Procedure: Awake Proning — The duration of proning will be a total of 8-10 hours with 1-2 hours break in supine position.
  Arms: Intervention - Awake Proning

SUMMARY:
The aim of the COVI-PRONE Trial is to determine if early awake prone positioning in COVID-19 patients with hypoxemic respiratory failure; irrespective of the mode of oxygen delivery; reduces the need for invasive mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years of age.
2. Suspected or confirmed COVID-19. Defined as: a positive PCR for SARS CoV-2 or pending PCR results for patients that are suspected to have COVID-19.
3. Hypoxemia on room air (SPO2<90%), and oxygen requirement ≥ 0.4 FiO2 (i.e. ≥ 40% oxygen).
4. Bilateral or unilateral chest infiltrates on x-ray as interpreted by the treating team.
5. Admitted to the ICU or an acute care bed where hemodynamic and respiratory monitoring is feasible.

Exclusion Criteria:

1. Immediate need for intubation as determined by the treating team.
2. Decreased level of consciousness (Glasgow Coma Scale score <10), or significant cognitive impairment hat may interfere with compliance (delirium, dementia)
3. Contraindication to proning including, but not limited to any of the following:

   Open chest or abdomen, abdominal surgery (i.e. laparotomy) within the 4 days, Unstable spine, facial, cervical, femur, or pelvic fractures. Limited neck mobility or inability to lie prone comfortably Skeletal deformities that interfere with proning. Complete bowel obstruction. Active upper gastrointestinal bleeding. Patient is unlikely/unable to prone, or to be compliant as indicated by the treating team.
4. Body mass index > 40 kg/m2
5. Pregnancy - third trimester.
6. Patient/substitute decision maker or caring physician's refusal to enroll in the study.
7. Patients with hemodynamic instability and moderate to high dose of vasopressors (norepinephrine dose ≥ 0.15 mcg/kg/min)
8. Intubation is not within patient's goals of care
9. Patient received awake proning session for > 1 day prior to randomization
10. Previous intubation within the same hospital admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2021-07-17 (Actual); Study Completion 2021-07-17 (Actual)

PRIMARY OUTCOMES:
Endotracheal intubation | within 30 days of randomization
  Medical procedure in which a tube is placed into the windpipe (trachea) through the mouth.

SECONDARY OUTCOMES:
Mortality | 60 days
  Death
Invasive mechanical ventilation free days | censored at 30 Days
  Number of days not receiving mechanical ventilation
Non-invasive ventilation free days | censored 30 days
  Number of days not receiving non-invasive mechanical ventilation
Days alive and outside ICU | 60 Days
  Number of days alive and outside the ICU
Days alive and outside of hospital | 60 days
  Number of days alive and outside of hospital
Complications from proning, | 30 days
  Includes any of the following: accidental removal of intravenous access, hypotension, pressure injuries, or other.

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Alhazzani, Principal Investigator — St. Joseph's Healthcare Hamilton; Yaseen Arabi, Principal Investigator — King Saud Bin Abdulaziz University for Health Sciences; Zainab Alduhailib, Principal Investigator — King Faisal Specialist Hospital and Research Center, Jeddah
Locations (17):
- University of Texas Health Sciences Centre, Dallas, Texas, United States
- Canada (8):
  - Univeristy of Calgary, Calgary, Alberta
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Hamilton General Hospital, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario
  - St. Catharine's General -, St. Catharines, Ontario
  - Sinai Health System, Toronto, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - CHU de Québec - Université Laval, Québec
- Kuwait (2):
  - Al-Amir Hospital, Kuwait City
  - Jaber Al Ahmed hospital, Kuwait City
- Saudi Arabia (6):
  - King Fahad Hospital of the University, Khobar, Eastern Province
  - Prince Mohammed bin Abdulaziz Hospital, Al Madīnah
  - King Abdulaziz Hospital - NGHA, AlAhsa
  - King Abdulaziz Medical City - Jeddah, Jeddah
  - King Abdulaziz Medical City, Riyadh
  - King Faisal Specialist Hospital & Research Center, Riyadh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alhazzani W, Parhar KKS, Weatherald J, Al Duhailib Z, Alshahrani M, Al-Fares A, Buabbas S, Cherian SV, Munshi L, Fan E, Al-Hameed F, Chalabi J, Rahmatullah AA, Duan E, Tsang JLY, Lewis K, Lauzier F, Centofanti J, Rochwerg B, Culgin S, Nelson K, Abdukahil SA, Fiest KM, Stelfox HT, Tlayjeh H, Meade MO, Perri D, Solverson K, Niven DJ, Lim R, Moller MH, Belley-Cote E, Thabane L, Tamim H, Cook DJ, Arabi YM; COVI-PRONE Trial Investigators and the Saudi Critical Care Trials Group. Effect of Awake Prone Positioning on Endotracheal Intubation in Patients With COVID-19 and Acute Respiratory Failure: A Randomized Clinical Trial. JAMA. 2022 Jun 7;327(21):2104-2113. doi: 10.1001/jama.2022.7993. PMID 35569448
- [Derived] Alhazzani W, Evans L, Alshamsi F, Moller MH, Ostermann M, Prescott HC, Arabi YM, Loeb M, Ng Gong M, Fan E, Oczkowski S, Levy MM, Derde L, Dzierba A, Du B, Machado F, Wunsch H, Crowther M, Cecconi M, Koh Y, Burry L, Chertow DS, Szczeklik W, Belley-Cote E, Greco M, Bala M, Zarychanski R, Kesecioglu J, McGeer A, Mermel L, Mammen MJ, Nainan Myatra S, Arrington A, Kleinpell R, Citerio G, Lewis K, Bridges E, Memish ZA, Hammond N, Hayden FG, Alshahrani M, Al Duhailib Z, Martin GS, Kaplan LJ, Coopersmith CM, Antonelli M, Rhodes A. Surviving Sepsis Campaign Guidelines on the Management of Adults With Coronavirus Disease 2019 (COVID-19) in the ICU: First Update. Crit Care Med. 2021 Mar 1;49(3):e219-e234. doi: 10.1097/CCM.0000000000004899. PMID 33555780